CLINICAL TRIAL: NCT00426920
Title: Evaluation of the Pharmacokinetics and Pharmacodynamics of Spray-Dried Recombinant Human Insulin Powder for Inhalation Administered Via a Dry Powder Inhalation Device Relative to SC Recombinant Human Insulin in Healthy Male Volunteers
Brief Title: Investigating the Pharmacokinetics and Pharmacodynamics of Recombinant Human Insulin Administered by Dry Powder Inhaler
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: QDose Limited (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IOV/QD001
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes Mellitus
Keywords: pharmacokinetics; pharmacodynamics; inhaled; recombinant human insulin
MeSH Terms: conditions — Diabetes Mellitus; Respiratory Aspiration | interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
Evaluation of the pharmacokinetics and pharmacodynamics of different doses of spray-dried recombinant human insulin powder for inhalation administered via a dry powder uinhalation device compared with subcutaneously administered regular human insulin in healthy male volunteers under the conditions of a eugycemic clamp.

DETAILED DESCRIPTION:
Explorative, single-center, randomized, open label, 4-way crossover study to evaluate the pharmacokinetics and pharmacodynamics of different doses of spray-dried recombinant human insulin powder for inhalation administered via a dry powder uinhalation device compared with subcutaneously administered regular human insulin in healthy male volunteers under the conditions of a eugycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* male
* non smoking for at least 12 months
* BMI equal to or less than 28
* no clinically significant abnormalities
* FVC and FEV1 equal to or more than 80%
* willing to participate and to sign informed consent form

Exclusion Criteria:

* positive results for insulin antibodies at screening
* history of substance abuse or dependency within last 5 years
* positive screening test for substance abuse
* positive blood test for HIV, hepatitis B or hepatitis C antibody
* fasting blood glucose of more than 126mg/dl
* any existing medical conditions which might interfere with absoprtion, distribution, metabolism or excretion of study medication
* history of bronchospastic disease(asthma), tachycardia, migraine headache, hypoglycemic episodes, jaundice, liver diseases, arterial hemorrhaging, severe hypertension or hypotension, cardiac abnormality, renal disease, allergies, unresolved psychiatric illness, drug-induced myopathy or any other clinically significant abnormality
* has received investigational medications within 21 days prior to receiving the first dose of study medication
* has taken or used any prescription medications within 21 days prior to receiving the first dose of study medication
* has taken or used any OTC medications,vitamins or herbal and/or nutritional supplements within 10 days days prior to receiving the first dose of study medication
* health that may be adversely affected by procedures or medications used in the study
* unwillingness or inability to understand or to follow required study restrictions and procedures

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2007-02

PRIMARY OUTCOMES:
maximum insulin serum concentration
early T50%
late T50%
Tmax
AUC

SECONDARY OUTCOMES:
maximum glucose infusion rate
early T50%
late T50%
Tmax
AUC

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, MD, Principal Investigator — Profil Institute for Clinical Research Incorporated
Locations (1):
- Profil Institute for Clinical Research Incorporated, Chula Vista, California, United States